CLINICAL TRIAL: NCT06184932
Title: TeleRehab to Restore Upper Limb Function in People With Chronic TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1217-23
Record Dates: First submitted 2023-07-05; First posted 2023-12-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury; Upper Extremity Dysfunction; Disability Physical
Keywords: upper limb; telerehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Arm and Hand Exercise (HAHE) (Experimental): An occupational therapist (OT) will incorporate participants' preference, goals, and current function to co-create UL exercise activities with participants. The exercise activities will be based on real-life activities that participants are familiar with. During the 6-week TeleRehab period, participants will complete 30 one-hour sessions of UL exercise activities, on their own without immediate supervision.
  Interventions: Behavioral: HAHE
- Exergame (Experimental): An occupational therapist (OT) will incorporate participants' preference, goals, and current function to select UL exercise activities with participants from the RehabKit program software. During the 6-week TeleRehab period, participants will complete 30 one-hour sessions of UL exercise activities, on their own without immediate supervision.
  Interventions: Behavioral: Exergame

INTERVENTIONS:
Behavioral: HAHE — Participants will self-initiate rehabilitative activities through the HAHE program.
  Arms: Home-based Arm and Hand Exercise (HAHE)
Behavioral: Exergame — Participants will self-initiate rehabilitative activities through the Exergame program.
  Arms: Exergame

SUMMARY:
The study aims to inform the subsequent large-scale clinical trial focused on using telerehabilitation techniques and technologies to improve upper limb function and quality of life.

DETAILED DESCRIPTION:
Upper limb (UL) function is often impaired and not fully recovered after moderate-to-severe traumatic brain injury (TBI), leading to devastating consequences and reducing quality of life. Clinicians have been encouraged to include UL rehabilitation, but existing evidence is insufficient to inform specific treatments for the TBI population. There is urgency to broaden the scientific evidence critical to advancing UL rehabilitation for TBI survivors, especially those living in the community with chronic UL impairment.

The study will examine two UL exercise programs through tele-rehabilitation (TeleRehab) techniques. Both programs are focused on functional tasks and daily activities. One program is implemented directly in the real-life home environment, the home-based arm and hand exercise (HAHE) program. The other program is delivered through simulated real-world scenarios, the exercise video game (Exergame) program. The HAHE program consists of UL exercises based on real-life activities that involve materials and objects readily available at home or easily obtained in regular stores. The Exergame program packages UL exercises into game-like activities delivered through a non-immersive virtual reality device.

Individuals with chronic UL impairment after moderate-to-severe TBI will participate in the proposed study. They will be randomly assigned to the HAHE or the Exergame program. Patients will complete 30 sessions of the assigned program over 6 weeks at home, with no immediate supervision. An occupational therapist will review the progress, assist in goal setting, and provide consultation to patients at the beginning of each week via a video call. The investigators will determine which of the programs is effective, and whether the programs lead to similar or different outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Time post injury > 12 months
* Moderate-to-severe TBI
* One upper limb (UL) is more affected than the other, and the participant reports impaired UL function because of the more affected limb.
* The more affected limb is at the Brunnstrom Stage 3, 4, or 5 of Arm Recovery .
* Meeting the following technology requirements: possessing and using a smartphone, Internet connection at home, and having a TV at home

Exclusion Criteria:

* < 18 years old at the time of injury
* A history of previous neurological disorder
* A history of substance abuse requiring inpatient treatment
* The more affected limb is at the Brunnstrom Stage 1, 2, 6, or 7 of Arm Recovery.
* Experiencing severe pain during the Brunnstrom Stage evaluation
* Active subluxation of the shoulders
* Living outside of the 50-mile radius of Kessler Foundation (West Orange, NJ)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Box and Block Test | 4 weeks before intervention, immediately before intervention, and immediately after intervention
  Participants will be seated at a table, face a rectangular box that is divided into two square compartments of equal dimensions on the left and right sides by means of a partition. At the beginning of the test, 150 1-inch blocks are in the same compartment. The task is to move as many blocks as possible, one at a time, from one compartment to the other using one arm only.
  Participants will be assessed 4 weeks before intervention (Time 1), immediately before (Time 2) and immediately after intervention (Time 3). The investigators will measure the change between Time 1 and Time 2 (baseline change), and the change between Time 2 and Time 3 (treatment change). The outcome measure is the difference between the two changes.
Wolf Motor Function Test | 4 weeks before intervention, immediately before intervention, and immediately after intervention
  The test quantitatively measures UL motor ability through 15 timed and functional tasks - forearm to table, forearm to box, extend elbow, extend elbow with weight, hand to table, hand to the box, reach and retrieve, lift can, lift pencil, lift paper clip, stack checkers, flip cards, turn key in lock, fold towel, and lift basket.
  Participants will be assessed 4 weeks before intervention (Time 1), immediately before (Time 2) and immediately after intervention (Time 3). The investigators will measure the change between Time 1 and Time 2 (baseline change), and the change between Time 2 and Time 3 (treatment change). The outcome measure is the difference between the two changes.

SECONDARY OUTCOMES:
Quality of Life in Neurological Disorders Measurement System | 4 weeks before intervention, immediately before intervention, and immediately after intervention
  The standardized short forms for adults evaluate anxiety, depression, fatigue, UL function, lower limb function, cognitive function, emotional and behavioral dyscontrol, positive affect and well-being, sleep disturbance, ability to participate in social roles and activities, satisfaction with social roles and activities, stigma, and communication.
  Participants will be assessed 4 weeks before intervention (Time 1), immediately before (Time 2) and immediately after intervention (Time 3). The investigators will measure the change between Time 1 and Time 2 (baseline change), and the change between Time 2 and Time 3 (treatment change). The outcome measure is the difference between the two changes.

CONTACTS AND LOCATIONS:
Overall Officials: Peii Chen, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States